CLINICAL TRIAL: NCT05390502
Title: Evaluation of a University of California-wide Quality Improvement Effort to Improve Blood Pressure Control Using Remote (Home) Monitoring
Brief Title: University of California Health Remote (Home) Monitoring Evaluation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of California, Los Angeles (Other)
Collaborators: University of California Office of the President- Quality and Population Health Management (Unknown); University of California, Davis (Other); University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Catherine A. Sarkisian, Director, Value-Based Care Research Consortium, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 22000036
Record Dates: First submitted 2022-05-20; First posted 2022-05-25 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Hypertension
Keywords: Remote Blood Pressure Monitoring
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Integrated (Experimental): Participants will have their home blood pressure readings sent directly to their participating health systems. Participants will also receive a wrap-around intervention.
  Interventions: Behavioral: integrated monitoring and local wrap-around hypertension program
- Manual (Active Comparator): Participants will record their own blood pressures and report them to their health care system as per usual care.
  Interventions: Behavioral: manual monitoring and general education on use

INTERVENTIONS:
Behavioral: manual monitoring and general education on use — Patients will receive a standard blood pressure monitor and education on how to use it. Data will be reported as part of usual care.
  Arms: Manual
Behavioral: integrated monitoring and local wrap-around hypertension program — Patients will receive a standard blood pressure monitor and a local wrap-around hypertension program. Data will be sent directly to their participating health system.
  Arms: Integrated

SUMMARY:
This study sets out to evaluate a University of California-wide (Davis, San Francisco, and Los Angeles) quality improvement initiative to increase remote (home) blood pressure monitoring and improve blood pressure control for persons with hypertension. Participants at each site will be randomized to one of two types of remote monitoring: integrated versus manual. Participants using the integrated monitoring will have their home blood pressure readings sent directly to their participating health systems. Participants using the manual monitoring will record their own blood pressures and report them to their health care system as per usual care.

DETAILED DESCRIPTION:
Hypertension is an important modifiable risk factor for numerous adverse health outcomes including cardiovascular and kidney disease. In 2017, about 45.3% of US adults had hypertension or were taking antihypertensive medications (1).

Hypertension has historically been diagnosed and treated using office-based blood pressure measurements, however blood pressure may differ when measured in the office compared to the home setting. Because of this discrepancy, and an extensive body of evidence supporting remote monitoring, national guidelines for hypertension management now recommend that all persons with hypertension participate in remote (home) monitoring. (2)

This study sets out to evaluate a University of California-wide (Davis, San Francisco, and Los Angeles) quality improvement initiative to increase remote (home) blood pressure monitoring and improve blood pressure control for persons with hypertension. Participants at each site will be randomized to one of two types of remote monitoring: integrated versus manual. Participants using the integrated monitoring will have their home blood pressure readings sent directly to their participating health systems. Participants using the manual monitoring will record their own blood pressures and report them to their health care system as per usual care.

The investigators hypothesize that remote monitoring (both integrated and manual) will be associated with improved blood pressure control and that there will be no difference in control between type of remote monitoring.

Aim 1: Evaluate whether this remote blood pressure quality improvement initiative leads to improved blood pressure control.

Aim 2: Compare the impact of integrated versus manual remote monitoring on blood pressure control.

The primary outcome measures will be: 1) the difference in blood pressure after six months (adjusted for baseline variables), and 2) whether participants achieved greater than or equal to 5 mmHg change in systolic blood pressure (SBP).

Outcomes will be compared between participants in each arm to determine whether one type of monitoring is superior to the other.

The investigators will convene bi-monthly meetings with site champions to foster communication and learning across sites and to learn about variation across sites.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years and older.
* Participant must be willing and functionally able (with help from another person if needed) to both use the remote BP monitoring device as well as do home BP monitoring using a manual BP cuff.
* Have access to the online healthcare portal (with help from another person if needed).

  •-Have outpatient visit within the last 12 months, and have a prior visit within 6 months of inclusion outpatient visit with diagnosis of hypertension, defined as having two readings of SBP > 140 or DBP > 90 mmHg
* Has visit with a primary care physician within one year.
* Takes zero or three anti-hypertensive prescriptions (can include pills with 2 different drugs so could be on 2 medications).

Exclusion Criteria:

* BP > 180/110 mmHg (office) or > 175/105 mmHg (self-measured BP measurements)
* Pheochromocytoma
* Uncontrolled hypothyroidism or hyperthyroidism
* Renal artery stenosis
* Conn's syndrome
* End stage renal disease (ESRD)
* Chronic kidney disease (CKD) Stage 3b (CrCL < 45) and above
* Transplant patients --> used the code that if they ever had a transplant
* Pregnancy
* Severe aortic stenosis
* Hospice/End-of-life or Palliative Care
* Left Ventricular Ejection Fraction < 30%
* Acute cardiac event in the last 3 months (e.g. acute MI)
* Heart block and arrhythmia(s)
* Recurrent or symptomatic hypotension (SBP < 100 mmHg or DBP < 60 mmHg)
* Drug/alcohol abuse
* Orthostatic hypotension (drop in SBP >20 mmHg)
* Other secondary causes of hypertension
* Receiving hypertension management from other services (home health, hospice, already enrolled in hypertension management program)
* White coat hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 660 (Estimated)
Dates: Start 2023-03-28 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Continuous change in blood pressure (BP) | Baseline, six months
  the difference in systolic blood pressure after six months (adjusted for baseline variables)

SECONDARY OUTCOMES:
Binary 5mm change in blood pressure | Baseline, six months
  whether participants achieved greater than or equal to 5 mmHg change in systolic blood pressure
Binary measure of controlled vs uncontrolled hypertension | Baseline, six months
  where uncontrolled is defined as SBP > 130 mmHg or diastolic blood pressure (DBP) > 80 mmHg.
Exploratory pre-post analysis of overall change in BP | Baseline, six months
  for all participants, subanalysis for select demographics including elderly.
Changes in blood pressure (BP) outcomes from integrated monitor readings | Baseline, six months
  For participants in the integrated device study arm, we will calculate the change between the baseline BP and the latest BP reading that is recorded via the remote device.

OTHER OUTCOMES:
Adverse events | Baseline, six months
  acute coronary syndrome, myocardial infarction, non-ST-elevation myocardial infarction (NSTEMI), ST Elevation Myocardial Infarction (STEMI), stroke (ischemic, hemorrhagic), decompensated heart failure, all-cause mortality, hospitalization, syncope, hyponatremia, hypokalemia, hyperkalemia

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Sarkisian, MD, MSHS, Principal Investigator — Director, Value-Based Care Research Consortium
Locations (3):
- United States (3):
  - University of California, Davis, Davis, California
  - University of California, Los Angeles, Los Angeles, California
  - University of California, San Francisco, San Francisco, California

REFERENCES:
- [Background] Carey RM, Whelton PK. The 2017 American College of Cardiology/American Heart Association Hypertension Guideline: A Resource for Practicing Clinicians. Ann Intern Med. 2018 Mar 6;168(5):359-360. doi: 10.7326/M18-0025. Epub 2018 Jan 23. No abstract available. PMID 29357396
- [Background] Shimbo D, Artinian NT, Basile JN, Krakoff LR, Margolis KL, Rakotz MK, Wozniak G; American Heart Association and the American Medical Association. Self-Measured Blood Pressure Monitoring at Home: A Joint Policy Statement From the American Heart Association and American Medical Association. Circulation. 2020 Jul 28;142(4):e42-e63. doi: 10.1161/CIR.0000000000000803. Epub 2020 Jun 22. PMID 32567342
- [Derived] Lee DR, Chenoweth M, Chuong LH, Villaflores CW, Cuevas M, Vangala S, Borenstein J, Kwak H, Chima-Melton C, Han M, Skootsky SA, Chan Tack T, Branagan L, Martin H, Gupta R, Phan L, Sanchez MA, Malaak MM, Dermenchyan A, Pearson KN, Altunyan M, Barakat PF, Pablo R, Sarkisian C. A Multisite Electronic Health Record Integrated Remote Monitoring Intervention for Hypertension Improvement: Protocol for a Randomized Pragmatic Comparative Effectiveness Trial. JMIR Res Protoc. 2023 Oct 30;12:e45915. doi: 10.2196/45915. PMID 37902819